CLINICAL TRIAL: NCT00100607
Title: Safety and Efficacy of AAE581 in Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE581A2203
Record Dates: First submitted 2005-01-03; First posted 2005-01-04 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Osteoporosis
Keywords: osteoporosis/osteopenia, BMD, postmenopausal
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic

INTERVENTIONS:
Drug: AAE581

SUMMARY:
This study will test the safety and efficacy of AAE581 in increasing Lumbar Spine bone mineral density (BMD) at 12 months, by Dexa-scan (DXA) in postmenopausal women with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* BMD T Score between -2 to -3.5
* 50-75 years old

Exclusion Criteria:

* Urolithiasis
* Bisphosphonates

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 676 (Actual)
Dates: Start 2004-02; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Lumbar spine BMD and total hip BMD after 1 year treatment
Safety and tolerability of one year treatment with different doses

SECONDARY OUTCOMES:
Effect of the different doses on BMD of lumbar spine, femoral neck, total hip, forearm and total body
Effect of the different doses on markers for bone formation and bone resorption
Structural information on cortical and trabecular bone at different anatomic sites after 6 and 12 months of treatment
Histological information on bone biopsy after 12 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals